CLINICAL TRIAL: NCT02148718
Title: Rapidity of Onset of Response to Adalimumab in Luminal Crohn's Disease (RAPIDA Study)
Brief Title: Rapidity of Response to Adalimumab Treatment in Patients With Crohn´s Disease
Acronym: RAPIDA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Laboratorio Echevarne (Industry); Pivotal S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W13-984; 2013-004781-34 (EudraCT Number)
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Results first posted 2017-08-29 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Moderate to Severe Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab (Experimental): Participants received adalimumab for 12 weeks (160 mg at Week 0; 80 mg at week 2; then adalimumab 40 mg every other week starting at Week 4).
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — Adalimumab pre-filled syringe, administered by subcutaneous injection
  Other Names: Humira, ABT-D2E7

SUMMARY:
The purpose of this study is to evaluate the rapidity of onset of clinical response to adalimumab therapy in patients with luminal Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease (CD) diagnosed within, at least, the previous 4 months.
* Patients with active luminal (Harvey-Bradshaw Index [HBI] ≥ 8) moderate to- severe CD.
* No response to a full and adequate course of therapy with a corticosteroid and/or an immunosuppressant.
* If receiving any of the following treatments, their dose should be stable during the periods indicated:

  * Aminosalicylates for, at least, the last 4 weeks
  * Probiotics for, at least, the last 4 weeks
  * Analgesics for, at least, the last 4 weeks
  * Antidiarrheals for, at least, the last 4 weeks
  * CD-related antibiotics for, at least, the last 4 weeks
  * Azathioprine, 6-mercaptopurine or methotrexate for, at least, the last 12 weeks
* If receiving any of the following treatments, their dose should not have been increase in the past two weeks (the dose reduction is permitted):

  * Oral budesonide (maximum dose of 9 mg/day)
  * Oral prednisone or equivalent (maximum dose of 40mg/day)

Exclusion Criteria:

* Previous treatment with any anti-Tumor Necrosis Factor agent
* Surgical bowel resection within the previous 6 months, ostomy, extensive bowel resection (> 100 cm), short bowel syndrome
* Fistulising Crohn's disease
* Treatment with cyclosporine or tacrolimus within the previous 8 weeks
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months from screening, congestive heart failure of worse than grade II New York criteria (New York Heart Association Functional Classification).
* Subject with an ostomy or ileoanal pouch, proctocolectomy, total colectomy, ileostomy, stoma or ileal pouch-anal anastomosis (Subjects with a previous ileo-rectal anastomosis are not excluded).
* Screening laboratory values (according to central laboratory)
* Known hepatitis C (HC) infection.
* Serologic evidence of hepatitis B (HB) infection based on the results of testing for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (anti-HBc) and hepatitis B surface antibody (anti-HBs) antibodies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Marín, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañon

REFERENCES:
- See also: Related info. — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 100 participants were enrolled in the study; 14 participants did not receive study drug and are excluded from the analyses.
Period: Overall Study
Arm/Group | Adalimumab
Started (Intent to Treat (ITT) population: all enrolled participants who received ≥ 1 dose of study drug) | 86
Completed | 55
Not Completed | 31
Not completed — Protocol Violation | 26
Not completed — Discontinued Study Prematurely | 5

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population: all enrolled participants who received at least 1 dose of study drug
Arm/Group | Adalimumab
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.73 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 37
Region of Enrollment [Number; unit: participants]
  Spain | 86

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Response at Day 4
Description: Clinical response defined as a decrease of at least 3 points in Harvey-Bradshaw Index (HBI) score. The HBI consists of only clinical parameters (general well-being, abdominal pain, number of liquid stools per day, abdominal mass, and complications): The first 3 items are scored for the previous day. Patients with Crohn's disease who scored 3 or less on the HBI are very likely to be in remission. Patients with a score of 8 to 9 or higher are considered to have severe disease.
Time Frame: Day 4
Population: Intent to Treat (ITT) population: all enrolled participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 86
percentage of participants | 61.63 [50.51 to 71.92]

2. Secondary Outcome: Percentage of Participants With Clinical Response at Week 1
Description: Clinical response defined as a decrease of at least 3 points in HBI score. The HBI consists of only clinical parameters (general well-being, abdominal pain, number of liquid stools per day, abdominal mass, and complications): The first 3 items are scored for the previous day. Patients with Crohn's disease who scored 3 or less on the HBI are very likely to be in remission. Patients with a score of 8 to 9 or higher are considered to have severe disease.
Time Frame: Week 1
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 86
percentage of participants | 75.58 [65.13 to 84.20]

3. Secondary Outcome: Percentage of Participants With Clinical Remission at Weeks 2 and 4
Description: Clinical remission defined as HBI < 5. The HBI consists of only clinical parameters (general well-being, abdominal pain, number of liquid stools per day, abdominal mass, and complications): The first 3 items are scored for the previous day. Patients with Crohn's disease who scored 3 or less on the HBI are very likely to be in remission. Patients with a score of 8 to 9 or higher are considered to have severe disease.
Time Frame: Weeks 2 and 4
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 86
percentage of participants
  Week 2 | 54.65 [43.55 to 65.42]
  Week 4 | 62.79 [51.70 to 72.98]

4. Secondary Outcome: European Quality of Life (EuroQol) 5 Dimensions 3 Levels Questionnaire (EQ-5D-3L) Index Score: Change From Baseline to Week 12
Description: The EQ-5D-3L is a standardized instrument for use as a measure of health-related quality of life (HRQoL) and consists of 2 components:
  1. The EQ-5D-3L Index Score has five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) with 3 levels of severity for each dimension ('no problems', 'some problems', and 'extreme problems'). The level of severity reported on each of the EQ-5D-3L dimensions determines a unique health state. Health states are converted into a weighted health state index. These weights lie on a scale on which full health has a value of 1 and dead has a value of 0.
  2. The EQ-5D visual analog scale (VAS) is a 20-cm scale with endpoints labeled "best imaginable health" and "worst imaginable health" anchored at 100 and 0, respectively.
  A positive change represents an improvement in HRQoL. Mean Baseline and mean change from Baseline to Week 12 in the EQ-5D-3L Index Score are presented.
Time Frame: Baseline (Week 0) and Week 12
Population: All participants in the ITT population with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
units on a scale
  Baseline | 0.62 (0.22)
  Change from Baseline to Week 12 | 0.14 (0.25)

5. Secondary Outcome: European Quality of Life (EuroQol) 5 Dimensions 3 Levels Questionnaire (EQ-5D-3L) Visual Analog Scale (VAS): Change From Baseline to Week 12
Description: The EQ-5D-3L is a standardized instrument for use as a measure of HRQoL and consists of 2 components:
  1. The EQ-5D-3L Index Score has five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) with 3 levels of severity for each dimension ('no problems', 'some problems', and 'extreme problems'). The level of severity reported on each of the EQ-5D-3L dimensions determines a unique health state. Health states are converted into a weighted health state index. These weights lie on a scale on which full health has a value of 1 and dead has a value of 0.
  2. The EQ-5D VAS is a 20-cm scale with endpoints labeled "best imaginable health" and "worst imaginable health" anchored at 100 and 0, respectively.
  A positive change represents an improvement in HRQoL. Mean Baseline and mean change from Baseline to Week 12 in the EQ-5D-3L VAS are presented.
Time Frame: Baseline (Week 0) and Week 12
Population: All participants in the ITT population with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 82
units on a scale
  Baseline | 55.36 (18.52)
  Change from Baseline to Week 12 | 15.37 (21.36)

6. Secondary Outcome: Inflammatory Bowel Disease Quality-36 (IBDQ-36) Questionnaire Overall Score: Change From Baseline to Week 12
Description: The IBDQ-36 is used to assess the HRQoL related to bowel symptoms. The IBDQ-36 overall score is calculated as the sum of thirty-six items, each scored on a 1 to 7 likert point scale, and ranges from 7 to 252. The highest score indicates the best HRQoL related to bowel symptoms. A positive change in IBDQ-36 overall score indicates an improvement in HRQoL due to inflammatory bowel disease. Mean Baseline and mean change from Baseline to Week 12 in the EQ-5D-3L VAS are presented.
Time Frame: Baseline (Week 0) and Week 12
Population: All participants in the ITT population with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 78
units on a scale
  Baseline | 145.1 (35.83)
  Change from Baseline to Week 12 | 44.72 (37.98)

7. Secondary Outcome: Fatigue Impact Scale for Daily Use (D-FIS): Change From Baseline to Week 12
Description: The D-FIS is used to measure the impact of fatigue on the daily lives of persons. The D-FIS overall score was calculated as the sum of eight items, each scored on a 0 to 4 point scale, and ranges from 0 to 32. A higher score indicates a higher impact of fatigue on daily life. A negative change in D-FIS Overall Score means an improvement in HRQoL due to fatigue. Mean Baseline and mean change from Baseline to Week 12 are presented.
Time Frame: Baseline (Week 0) and Week 12
Population: All participants in the ITT population with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 79
units on a scale
  Baseline | 14.45 (8.53)
  Change from Baseline to Week 12 | -4.69 (8.44)

8. Secondary Outcome: Change From Baseline to Week 12 in Analytic Markers of Inflammation: Hemoglobin
Description: Analytic markers of inflammation are hemogram (hemoglobin, hematocrit, leukocytes, neutrophils, lymphocytes, monocytes, eosinophils, basophils, and platelets), erythrocytes sedimentation rate (ESR), C-reactive protein (CRP), fecal calprotectin, and coagulation (activated partial thromboplastin time [aPTT], international normalized ratio [INR], and fibrinogen). Mean Baseline and mean change from Baseline to Week 12 are presented.
Time Frame: Baseline (Week 0) and Week 12
Population: All participants in the ITT population with evaluable data
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Adalimumab
Number analyzed (Participants) | 84
g/dL
  Baseline | 13.01 (1.40)
  Change from Baseline to Week 12: number analyzed (Participants) | 79
  Change from Baseline to Week 12 | 0.27 (0.97)

9. Secondary Outcome: Change From Baseline to Week 12 in Analytic Markers of Inflammation: Hematocrit
Description: Analytic markers of inflammation are hemogram (hemoglobin, hematocrit, leukocytes, neutrophils, lymphocytes, monocytes, eosinophils, basophils, and platelets), erythrocytes, ESR, CRP, fecal calprotectin, and coagulation (aPTT, INR, and fibrinogen). Mean Baseline and mean change from Baseline to Week 12 for each parameter are presented.
Time Frame: Baseline (Week 0) and Week 12
Population: All participants in the ITT population with evaluable data
Measure: Mean (Standard Deviation); unit: % volume
Arm/Group | Adalimumab
Number analyzed (Participants) | 84
% volume
  Baseline | 39.47 (3.99)
  Change from Baseline to Week 12: number analyzed (Participants) | 79
  Change from Baseline to Week 12 | 0.86 (2.79)

10. Secondary Outcome: Change From Baseline to Week 12 in Analytic Markers of Inflammation: Leukocytes, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils, and Platelets
Description: as for outcome 9
Time Frame: Baseline (Week 0) and Week 12
Population: All participants in the ITT population with evaluable data
Measure: Mean (Standard Deviation); unit: cellsx10^3/uL
Arm/Group | Adalimumab
Number analyzed (Participants) | 84
cellsx10^3/uL
  Leukocytes Baseline | 8.11 (3.23)
  Leukocytes Change from Baseline to Week 12: number analyzed (Participants) | 79
  Leukocytes Change from Baseline to Week 12 | -1.62 (2.87)
  Neutrophils Baseline | 5.61 (2.86)
  Neutrophils Change from Baseline to Week 12: number analyzed (Participants) | 79
  Neutrophils Change from Baseline to Week 12 | -1.99 (2.87)
  Lymphocytes Baseline | 1.80 (0.94)
  Lymphocytes Change from Baseline to Week 12: number analyzed (Participants) | 79
  Lymphocytes Change from Baseline to Week 12 | 0.39 (0.76)
  Monocytes Baseline | 0.50 (0.25)
  Monocytes Change from Baseline to Week 12: number analyzed (Participants) | 79
  Monocytes Change from Baseline to Week 12 | -0.009 (0.219)
  Eosinophils Baseline | 0.17 (0.15)
  Eosinophils Change from Baseline to Week 12: number analyzed (Participants) | 79
  Eosinophils Change from Baseline to Week 12 | -0.010 (0.095)
  Basophils Baseline | 0.02 (0.02)
  Basophils Change from Baseline to Week 12: number analyzed (Participants) | 79
  Basophils Change from Baseline to Week 12 | 0.003 (0.033)
  Platelets Baseline | 316.1 (90.1)
  Platelets Change from Baseline to Week 12: number analyzed (Participants) | 79
  Platelets Change from Baseline to Week 12 | -40.4 (76.4)

11. Secondary Outcome: Change From Baseline to Week 12 in Analytic Markers of Inflammation: Erythrocytes
Description: as for outcome 9
Time Frame: Baseline (Week 0) and Week 12
Population: All participants in the ITT population with evaluable data
Measure: Mean (Standard Deviation); unit: cellsx10^6/uL
Arm/Group | Adalimumab
Number analyzed (Participants) | 84
cellsx10^6/uL
  Baseline | 4.37 (0.51)
  Change from Baseline to Week 12: number analyzed (Participants) | 79
  Change from Baseline to Week 12 | 0.052 (0.308)

12. Secondary Outcome: Change From Baseline to Week 12 in Analytic Markers of Inflammation: Sedimentation Rate (ESR)
Description: as for outcome 9
Time Frame: Baseline (Week 0) and Week 12
Population: All participants in the ITT population with evaluable data
Measure: Mean (Standard Deviation); unit: mm/1h
Arm/Group | Adalimumab
Number analyzed (Participants) | 84
mm/1h
  Baseline | 19.49 (18.38)
  Change from Baseline to Week 12: number analyzed (Participants) | 79
  Change from Baseline to Week 12 | -7.48 (14.26)

13. Secondary Outcome: Change From Baseline to Week 12 in Analytic Markers of Inflammation: C-reactive Protein (CRP)
Description: as for outcome 9
Time Frame: Baseline (Week 0) and Week 12
Population: All participants in the ITT population with evaluable data
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Adalimumab
Number analyzed (Participants) | 85
U/L
  Baseline | 11.06 (16.2)
  Change from Baseline to Week 12: number analyzed (Participants) | 80
  Change from Baseline to Week 12 | -7.61 (16.4)

14. Secondary Outcome: Change From Baseline to Week 12 in Analytic Markers of Inflammation: Fecal Calprotectin
Description: as for outcome 9
Time Frame: Baseline (Week 0) and Week 12
Population: All participants in the ITT population with evaluable data
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Adalimumab
Number analyzed (Participants) | 74
mg/kg
  Baseline | 1,550.4 (2,798.4)
  Change from Baseline to Week 12: number analyzed (Participants) | 61
  Change from Baseline to Week 12 | -1,043.8 (2,895.3)

15. Secondary Outcome: Change From Baseline to Week 12 in Analytic Markers of Inflammation: Activated Partial Thromboplastin Time (aPTT)
Description: as for outcome 9
Time Frame: Baseline (Week 0) and Week 12
Population: All participants in the ITT population with evaluable data
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Adalimumab
Number analyzed (Participants) | 85
sec
  Baseline | 30.58 (3.89)
  Change from Baseline to Week 12: number analyzed (Participants) | 79
  Change from Baseline to Week 12 | 0.76 (3.97)

16. Secondary Outcome: Change From Baseline to Week 12 in Analytic Markers of Inflammation: International Normalized Ratio (INR)
Description: as for outcome 9
Time Frame: Baseline (Week 0) and Week 12
Population: All participants in the ITT population with evaluable data
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Adalimumab
Number analyzed (Participants) | 85
ratio
  Baseline | 1.05 (0.06)
  Change from Baseline to Week 12: number analyzed (Participants) | 79
  Change from Baseline to Week 12 | 0.02 (0.07)

17. Secondary Outcome: Change From Baseline to Week 12 in Analytic Markers of Inflammation: Fibrinogen
Description: as for outcome 9
Time Frame: Baseline (Week 0) and Week 12
Population: All participants in the ITT population with evaluable data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Adalimumab
Number analyzed (Participants) | 85
mg/dL
  Baseline | 374.5 (68.17)
  Change from Baseline to Week 12: number analyzed (Participants) | 79
  Change from Baseline to Week 12 | -43.6 (65.7)

18. Secondary Outcome: Percentage of Participants With Clinical Response at Day 4 or Week 12 and Clinical Remission at Week 12
Description: The percentage of participants with clinical response (defined as decrease of at least 3 points in HBI score) at Day 4 or Week 1 and clinical remission (defined as a HBI < 5) at Week 12.
Time Frame: Up to Week 12
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 86
percentage of participants | 58.90

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until 70 days after the last dose of study drug (up to 20 weeks).
Description: TEAEs and TESAEs are defined as any AE or SAE with an onset date after the first dose of study drug until 70 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Adalimumab
Serious Adverse Events (participants affected / at risk) | 2/86
Other Adverse Events (participants affected / at risk) | 35/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=86)
Crohn's disease (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Pneumonia (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=86)
Anaemia (Blood and lymphatic system disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Eyelid disorder (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Presbyopia (Eye disorders) | 1
Abdominal mass (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 3
Aphthous ulcer (Gastrointestinal disorders) | 2
Crohn's disease (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Asthenia (General disorders) | 2
Fatigue (General disorders) | 1
General physical health deterioration (General disorders) | 1
Pyrexia (General disorders) | 2
Drug hypersensitivity (Immune system disorders) | 1
Cellulitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 3
Influenza (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 3
Pharyngotonsillitis (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 2
Rotavirus infection (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Blood triglycerides increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Weight decreased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.